CLINICAL TRIAL: NCT01569074
Title: (OSKIRA-Asia-1): A Multi-centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Dose Ranging Study in Asia Evaluating Efficacy and Safety of Fostamatinib in Patients With Active Rheumatoid Arthritis Who Are Inadequate Responders to Methotrexate Therapy
Brief Title: Evaluation of Safety and Effectiveness of Fostamatinib Compared to Placebo in Patients in Asia With Rheumatoid Arthritis
Acronym: OSKIRA-Asia-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: AZ decision to discontinue fostamatinib development in RA; rights to fostamatinib returned to Rigel Pharmaceuticals.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4300C00008
Record Dates: First submitted 2012-03-30; First posted 2012-04-02 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Dosing A regimen (Experimental): Oral treatment
  Interventions: Drug: Fostamatinib
- Dosing B regimen (Experimental): Oral treatment
  Interventions: Drug: Fostamatinib
- Dosing C regimen (Experimental): Oral treatment
  Interventions: Drug: Fostamatinib
- Dosign D regimen (Experimental): Oral treatment
  Interventions: Drug: Fostamatinib
- Dosing E regimen (Placebo Comparator): Oral treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib 100mg twice daily for 12 weeks
  Arms: Dosing A regimen
Drug: Fostamatinib — Fostamatinib 100mg twice daily for 4 weeks, followed by150mg once daily up to Week 12
  Arms: Dosing B regimen
Drug: Fostamatinib — Fostamatinib 75mg twice daily for 12 weeks
  Arms: Dosing C regimen
Drug: Fostamatinib — Fostamatinib 50mg twice daily for 12 weeks
  Arms: Dosign D regimen
Drug: Placebo — Placebo twice daily for 12 weeks
  Arms: Dosing E regimen

SUMMARY:
The purpose of the study is to evaluate the effectiveness of four dosing regimens of fostamatinib compared to placebo, in patients with rheumatoid arthritis (RA) who are taking methotrexate but not responding. The study will last for 12 weeks.

DETAILED DESCRIPTION:
(OSKIRA-Asia-1): A Multi-centre, Randomised, Double-Blind, Placebo-Controlled, Parallel Group Dose Ranging Study in Asia Evaluating Efficacy and Safety of Fostamatinib in Patients with Active Rheumatoid Arthritis who are Inadequate Responders to Methotrexate Therapy

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over
* Active rheumatoid arthritis (RA) diagnosed after the age of 16
* 6 or more swollen joints and 6 or more tender/painful joints from certain joints in the hands, wrists, arms and knees
* At least one of: positive result for rheumatoid factor test, either in the past or currently (blood test); x-ray showing bone erosion within the last 12 months; presence of certain antibodies in the blood (blood test)
* Currently taking methotrexate for at least 4 months (and on a stable dose for at least 6 weeks)

Exclusion Criteria:

* Females who are pregnant or breast feeding
* Certain inflammatory conditions (other than rheumatoid arthritis), connective tissue diseases or chronic pain disorders.
* Previously taken, but not responded to, certain biological treatments for rheumatoid arthritis
* High blood pressure that is not controlled by medication
* Low levels of neutrophils in the blood (blood test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil - Mackillop, MD, Study Director — AstraZeneca
Locations (34):
- Hong Kong (2):
  - Research Site, New Territories, HK
  - Research Site, Hong Kong
- Japan (20):
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kitakyushu-shi, Fukuoka
  - Research Site, Kurume, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kato-shi, Hyōgo
  - Research Site, Kasama-shi, Ibaraki
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Sendai, Miyagi
  - Research Site, Isahaya, Nagasaki
  - Research Site, Nagasaki, Nagasaki
  - Research Site, Omura-shi, Nagasaki
  - Research Site, Sasebo-shi, Nagasaki
  - Research Site, Shibata, Niigata
  - Research Site, Okayama, Okayama-ken
  - Research Site, Tomigusuku-shi, Okinawa
  - Research Site, Matsue, Shimane
  - Research Site, Hamamatsu, Shizuoka
  - Research Site, Shinjuku, Tokyo
  - Research Site, tabashi City, Tokyo
- South Korea (4):
  - Research Site, Anyang-si, Gyeonggi-do
  - Research Site, Gwangju
  - Research Site, Incheon
  - Research Site, Seoul
- Taiwan (4):
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (2):
  - Research Site, Bangkok
  - Research Site, Singapore
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

REFERENCES:
- [Derived] Tanaka Y, Millson D, Iwata S, Nakayamada S. Safety and efficacy of fostamatinib in rheumatoid arthritis patients with an inadequate response to methotrexate in phase II OSKIRA-ASIA-1 and OSKIRA-ASIA-1X study. Rheumatology (Oxford). 2021 Jun 18;60(6):2884-2895. doi: 10.1093/rheumatology/keaa732. PMID 33254235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 298 patients were enrolled: 31, 33, 33, 33 & 33 were randomised to Groups A, B, C, D & E respectively (all received at least 1 dose of investigational product).
Pre-assignment Details: A total of 135 patients failed screening.
Groups:
- FOSTA 100 MG BID PO: Dosing Group A
- FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO: Dosing Group B
- FOSTA 75 MG BID PO: Dosing Group C
- FOSTA 50 MG BID PO: Dosing Group D
- PLACEBO PO: Dosing Group E
Period: Overall Study
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Started | 31 (Patients who received treatment) | 33 (Patients who received treatment) | 33 (Patients who received treatment) | 33 (Patients who received treatment) | 33 (Patients who received treatment)
Randomised But Did Not Receive Treatment | 0 | 0 | 0 | 0 | 0
Completed | 24 (Number of patients who completed treatment includes patients who had a dose reduction.) | 24 (Number of patients who completed treatment includes patients who had a dose reduction.) | 21 (Number of patients who completed treatment includes patients who had a dose reduction.) | 25 (Number of patients who completed treatment includes patients who had a dose reduction.) | 25 (Number of patients who completed treatment includes patients who had a dose reduction.)
Not Completed | 7 | 9 | 12 | 8 | 8
Not completed — Study stopped | 6 | 6 | 8 | 7 | 7
Not completed — Study-specific discontinuation criteria | 0 | 1 | 0 | 0 | 0
Not completed — Severe non-compliance to protocol | 0 | 0 | 1 | 0 | 0
Not completed — eg change in circumstances | 0 | 2 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO | Total
Number analyzed (Participants) | 31 | 33 | 33 | 33 | 33 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14.3) | 55 (10.4) | 56 (11.5) | 50 (11.4) | 53 (11.3) | 53 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 27 | 31 | 28 | 142
  Male | 0 | 8 | 6 | 2 | 5 | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 31 | 33 | 33 | 33 | 33 | 163
  White | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Indian or Pakistani | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving ACR20 at Week 12, Comparison Between Fostamatinib and Placebo
Description: ACR20: American College of Rheumatology 20% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as C-Reactive Protein) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: 12 weeks
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle.
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 26 | 29 | 27 | 28 | 28
Percentage of responders | 53.8 | 55.2 | 25.9 | 46.4 | 32.1
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; Non-responder imputation has been applied following premature withdrawal, or increased dose of methotrexate or any DMARD initiation, or following receipt of any parenteral steroids, or for patients with no post baseline data. Subjects who prematurely withdrew due to project closure have no imputation applied; Test type: Superiority or Other; p = 0.059, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.23, 80% CI 2-sided [0.07 to 0.39]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.054, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.24, 80% CI 2-sided [0.08 to 0.39]
Statistical Analysis 3: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.570, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = -0.06, 80% CI 2-sided [-0.20 to 0.08]
Statistical Analysis 4: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.262, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.14, 80% CI 2-sided [-0.02 to 0.29]

2. Secondary Outcome: Proportion of Patients Achieving ACR20 at Week 1, Comparison Between Fostamatinib and Placebo
Description: ACR20: American College of Rheumatology 20% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as C-Reactive Protein) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally.
Time Frame: 1 week
Population: The full analysis set includes those patients who received at least 1 dose of investigational product. Patients were analysed by randomised treatment in accordance with the intention to treat principle. The fostamatinib 100 mg BID combined group contains 31 patients from Dosing Group A and 33 patients from Dosing Group B.
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO | FOSTA 100 MG BID PO
Number analyzed (Participants) | 33 | 33 | 33 | 64
Percentage of responders | 21.2 | 18.2 | 15.2 | 25.0
Statistical Analysis 1: Comparison: PLACEBO PO vs FOSTA 100 MG BID PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.172, Mantel Haenszel — Week 1; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.11, 80% CI 2-sided [0.01 to 0.21]
Statistical Analysis 2: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.489, Mantel Haenszel — Week 1; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.06, 80% CI 2-sided [-0.05 to 0.18]
Statistical Analysis 3: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.704, Mantel Haenszel — Week 1; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.03, 80% CI 2-sided [-0.08 to 0.15]

3. Secondary Outcome: Proportion of Patients Achieving ACR50 at Week 12, Comparison Between Fostamatinib and Placebo
Description: ACR50: American College of Rheumatology 50% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as C-Reactive Protein) and the physician and patient's own assessments of disease activity, pain and physical function, BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 26 | 29 | 27 | 28 | 28
Percentage of responders | 30.8 | 34.5 | 7.4 | 10.7 | 14.3
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.114, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.17, 80% CI 2-sided [0.03 to 0.31]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.035, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.21, 80% CI 2-sided [0.08 to 0.34]
Statistical Analysis 3: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.334, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = -0.07, 80% CI 2-sided [-0.17 to 0.02]
Statistical Analysis 4: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.645, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = -0.04, 80% CI 2-sided [-0.13 to 0.06]

4. Secondary Outcome: Proportion of Patients Achieving ACR70 at Week 12, Comparison Between Fostamatinib and Placebo
Description: ACR70: American College of Rheumatology 70% response criteria, based on count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (such as C-Reactive Protein) and the physician and patient's own assessments of disease activity, pain and physical function. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 26 | 29 | 27 | 28 | 28
Percentage of responders | 11.5 | 13.8 | 0 | 0 | 0
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.028, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.12, 80% CI 2-sided [0.05 to 0.19]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.021, Mantel Haenszel — Week 12; Treatment difference in proportion of responders, with a Mantel-Haenszel approach stratified by pooled country; Weighted difference in proportions = 0.14, 80% CI 2-sided [0.06 to 0.22]

5. Secondary Outcome: ACRn - Comparison Between Fostamatinib and Placebo at Week 12
Description: ACRn: American College of Rheumatology index of RA improvement, based on smallest percentage improvement in the count of swollen joints (out of 28 joints), count of tender joints (out of 28 joints), or in blood test measures of inflammation (such as C-Reactive Protein) or the physician or patient's own assessments of disease activity, pain and physical function. Scores are reported as a percentage improvement on a scale of -100 to +100, with larger values representing a better clinical outcome. Mean refers to change at Week 12. BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage improvement from baseline
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 26 | 29 | 27 | 28 | 28
Percentage improvement from baseline | 25.52 (37.029) | 24.18 (39.925) | 3.59 (29.774) | 15.88 (24.354) | 10.94 (28.302)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.073, Van Elteren — As this is a non-parametric test, p-values alone are presented rather than an estimated treatment difference; P-value estimated using the Van Elteren method stratified by pooled country
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.065, Van Elteren — As this is a non-parametric test, p-values alone are presented rather than an estimated treatment difference; P-value estimated using the Van Elteren test stratified by pooled country
Statistical Analysis 3: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.317, Van Elteren — As this is a non-parametric test, p-values alone are presented rather than an estimated treatment difference; P-value estimated using the Van Elteren method stratified by pooled country
Statistical Analysis 4: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.263, Van Elteren — As this is a non-parametric test, p-values alone are presented rather than an estimated treatment difference; P-value estimated using the Van Elteren method stratified by pooled country

6. Secondary Outcome: Proportion of Patients Achieving DAS28-CRP<=3.2 at Week 12, Comparison Between Fostamatinib and Placebo
Description: DAS28-CRP: Disease Activity Score based on a count of swollen and tender joints (out of 28 joints), blood test measures of inflammation (CRP) and the patient's own assessment. Scores can take any positive value with a lower value indicating a better clinical condition. DAS28-CRP score of <=3.2 indicates low disease activity. BID = twice daily, CRP = C-reactive protein, , DMARD = disease modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once daily.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 26 | 29 | 27 | 28 | 28
Percentage of responders | 34.6 (0.81) | 34.5 (0.82) | 22.2 (0.77) | 17.9 (0.75) | 10.7
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.033, Regression, Logistic; Odds ratio and 80% confidence intervals are calculated using Logistic Regression with treatment and pooled country as factors; Odds Ratio (OR) = 5.3, 80% CI 2-sided [1.94 to 14.31] — An odds ratio of >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.033, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 5.1, 80% CI 2-sided [1.92 to 13.61] — An odds ratio of >1 indicates a benefit towards fostamatinib
Statistical Analysis 3: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.257, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 2.5, 80% CI 2-sided [0.89 to 6.89] — An odds ratio of >1 indicates a benefit towards fostamatinib
Statistical Analysis 4: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.481, Regression, Logistic; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 1.8, 80% CI 2-sided [0.63 to 5.04] — An odds ratio of >1 indicates a benefit towards fostamatinib

7. Secondary Outcome: Proportion of Patients With DAS28-CRP EULAR Response at Week 12, Comparison Between Fostamatinib and Placebo
Description: Change from baseline in DAS28-CRP at Week 12 was derived and categorised using the European League Against Rheumatism (EULAR) response criteria. BID = twice a day, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once a day.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 26 | 29 | 27 | 28 | 28
Percentage of responders
  No response | 30.8 (1.46) [0.20 to 0.68] | 41.4 (1.34) [0.26 to 0.89] | 48.1 (1.30) [0.20 to 0.65] | 17.9 (1.58) | 35.7
  Moderate response | 34.6 | 24.1 | 29.6 | 64.3 | 53.6
  Good response | 34.6 | 34.5 | 22.2 | 17.9 | 10.7
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.131, Proportional odds model; No response, moderate response and good response are included in the proportional odds model with treatment and pooled country as factors; Odds Ratio (OR) = 2.17, 80% CI 2-sided [1.12 to 4.20] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.423, Proportional odds model; [statistical method as in outcome 7, analysis 1]; Odds Ratio (OR) = 1.49, 80% CI 2-sided [0.79 to 2.82] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 3: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.781, Proportional odds model; No response, moderate response and good response are included in the proportional odds model with treatment and country as factors; Odds Ratio (OR) = 0.87, 80% CI 2-sided [0.45 to 1.67] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 4: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.239, Proportional odds model; [statistical method as in outcome 7, analysis 3]; Odds Ratio (OR) = 1.81, 80% CI 2-sided [0.95 to 3.44] — An odds ratio >1 indicates a benefit towards fostamatinib

8. Secondary Outcome: Proportion of Patients With HAQ-DI Response at Week 12, Comparison Between Fostamatinib and Placebo
Description: HAQ-DI: Health Assessment Questionnaire - Disability Index, a measure of physical function. The HAQ-DI score is calculated by summing scores from 8 sub-categories (ie, scores for patient ability in dressing and grooming, rising, eating, walking, hygiene, reach, grip and common daily activities) and dividing by the number of categories completed. The HAQ-DI score takes values between 0 and 3, with higher score indicating greater disability. HAQ-DI response is a reduction from baseline in HAQ-DI greater than or equal to the minimally important difference (0.22). BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, OR = odds ratio, PO = orally, QD = once a day.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of responders
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 26 | 29 | 27 | 28 | 28
Percentage of responders | 69.2 | 48.3 | 44.4 | 46.4 | 50.0
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.169, Regression, Logistic — Week 12; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 2.2, 80% CI 2-sided [1.06 to 4.67] — An odds ration >1 indicates a benefit towards fostamatinib
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.833, Regression, Logistic — Week 12; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.9, 80% CI 2-sided [0.45 to 1.78] — An odds ratio >1 indicates a benefit towards fostamatinib
Statistical Analysis 3: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.614, Regression, Logistic — Week 12; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.8, 80% CI 2-sided [0.37 to 1.54] — An odds ratio of >1 indicates a benefit towards fostamatinib
Statistical Analysis 4: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.748, Regression, Logistic — Week 12; [statistical method as in outcome 6, analysis 1]; Odds Ratio (OR) = 0.8, 80% CI 2-sided [0.42 to 1.69] — An odds ratio of >1 indicates a benefit towards fostamatinib

9. Secondary Outcome: SF-36 - Comparison of the Change in PCS From Baseline Between Fostamatinib and Placebo at Week 12
Description: SF-36 = 36-item Short Form Health Survey, as a measure of health related quality of life. Scores for 8 sub-domains (Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Function, Role-Emotional and Mental Health) are derived and normalised to a scale of 0 to 100. The physical and mental component scores (PCS and MCS) are derived by multiplying each of these 8 scores by a constant, summing them and standardising against a population with mean of 50, standard deviation of 10. A higher score represents better quality of life. Mean changes from baseline are presented as increases from baseline (defined as post-baseline minus baseline); larger changes indicate a better clinical condition. Mean refers to change in scores at Week 12. ANCOVA = analysis of covariance, BID = twice daily, DMARD = disease-modifying anti-rheumatic drug, PO = orally, QD = once a day.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 25 | 29 | 26 | 27 | 27
Units on a scale | 7 (7.5) | 4 (7.4) | 3 (6.8) | 5 (5.6) | 3 (5.1)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.087, ANCOVA; Including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 3.01, 80% CI 2-sided [0.76 to 5.26]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.881, ANCOVA; Including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 0.25, 80% CI 2-sided [-1.91 to 2.41]
Statistical Analysis 3: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.806, ANCOVA; Includes terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = -0.42, 80% CI 2-sided [-2.64 to 1.80]
Statistical Analysis 4: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.548, ANCOVA; Includes terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 1.03, 80% CI 2-sided [-1.17 to 3.23]

10. Secondary Outcome: SF-36 - Comparison of the Change in MCS From Baseline Between Fostamatinib and Placebo at Week 12
Description: as for outcome 9
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 75 MG BID PO | FOSTA 50 MG BID PO | PLACEBO PO
Number analyzed (Participants) | 25 | 29 | 26 | 27 | 27
Units on a scale | 7 (8.7) | 6 (7.7) | 2 (7.0) | 5 (8.9) | 4 (7.9)
Statistical Analysis 1: Comparison: FOSTA 100 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.139, ANCOVA; Including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 3.12, 80% CI 2-sided [0.42 to 5.82]
Statistical Analysis 2: Comparison: FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.223, ANCOVA; Including terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 2.47, 80% CI 2-sided [-0.13 to 5.07]
Statistical Analysis 3: Comparison: FOSTA 75 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.432, ANCOVA; Includes terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = -1.63, 80% CI 2-sided [-4.30 to 1.04]
Statistical Analysis 4: Comparison: FOSTA 50 MG BID PO vs PLACEBO PO; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.481, ANCOVA; Includes terms for baseline as a continuous covariate and treatment and pooled country as factors; Treatment difference = 1.45, 80% CI 2-sided [-1.19 to 4.09]

ADVERSE EVENTS:
Arm/Group | FOSTA 100 MG BID PO | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO | FOSTA 50 MG BID PO | FOSTA 75 MG BID PO | PLACEBO PO
Serious Adverse Events (participants affected / at risk) | 1/31 | 1/33 | 3/33 | 0/33 | 1/33
Other Adverse Events (participants affected / at risk) | 21/31 | 17/33 | 17/33 | 16/33 | 15/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID PO (N=31) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO (N=33) | FOSTA 50 MG BID PO (N=33) | FOSTA 75 MG BID PO (N=33) | PLACEBO PO (N=33)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LARYNGITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FOSTA 100 MG BID PO (N=31) | FOSTA 100 MG BID (4 WKS) THEN 150 MG QD PO (N=33) | FOSTA 50 MG BID PO (N=33) | FOSTA 75 MG BID PO (N=33) | PLACEBO PO (N=33)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (3)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (6) | 2 (2) | 5 (7) | 4 (4) | 3 (5)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 5 (6) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (2) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
VOMITING (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
HEADACHE (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPERTENSION (Vascular disorders) | 8 (8) | 6 (6) | 3 (3) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days